CLINICAL TRIAL: NCT01227174
Title: Safety and Efficacy of Propofol Only Sedation in Oral and Maxillofacial Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atlantic Center for Oral and Maxillofacial Surgery (Other)
Responsible Party: Dr. Ben Davis, Atlantic Centre for Oral and Maxillofacial Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDHA-RS/2011-142
Record Dates: First submitted 2010-10-16; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Procedural Sedation; Propofol
Keywords: propofol only; safety and efficacy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol sedation (Experimental): Patients will be undergo procedural sedation using propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Procedural sedation will be achieved using propofol
  Other Names: Diprivan

SUMMARY:
The purpose of this study is to determine if the use of propofol only to achieve procedural sedation for the removal of third molars is both safe and effective.

DETAILED DESCRIPTION:
Removal of third molars is a common procedure performed in North America. Many surgeon choose to complete the procedure using procedural sedation. The most commonly used combination of medications to achieve procedural sedation consists of midazolam, fentanyl, and propofol. Propofol has been gaining increasing attention as a sedative agent due to its predictable pharmacokinetics and favorable amnestic properties. These properties make propofol an attractive sedative agent when compared to the benzodiazepines which are known to have a slower onset coupled with a much longer offset resulting in a prolonged sedative effect well beyond that required for completion of the procedure. Several studies have compared the use of propofol in combination with other sedatives with various control groups. These studies reliably confirm both the safety and efficacy of propofol. Some researches have speculated that the differences in nausea and vomiting reported by patients are secondary to the differences in dosage of fentanyl between groups. Others have concluded that fentanyl provides no advantage when using intermittent propofol in short duration procedures. Recent studies have found favourable results when using propofol only to achieve procedural sedation. On review of the Oral and Maxillofacial Surgery literature regarding this topic, a lack of internally and externally validated research was discovered. Oral and Maxillofacial surgical procedures are unique in duration of procedure and use of local anesthesia making it difficult to generalize data obtained from other specialties.

All eligible patients will be assigned to a single group. They will be asked to fill out a survey to determine their level of anxiety prior to the procedure. Participants will then proceed the same as non-study patients to see the nurse for a pre-operative assessment. After seeing the nurse, patients will see the surgeon for the procedure. Most of the data (blood pressure, heart rate, breathing rate etc.) is collected during the procedure. During procedural sedation monitoring is performed as usual but study patients will have capnometry added to the standard of care. Capnometry is a way of examining your breathing. It is the measurement of the carbon dioxide in the air that you breathe out through you nose. After the procedure is complete patients are transported to recovery where they must remain for a minimum of 30 minutes prior to discharge. The nurse in recovery will monitor you recovery continuously during your stay. The nurse will also apply a standard recovery score to your recovery every 5 minutes to track your progression. Once you are recovered from the procedural sedation you will be asked to complete a short questionnaire about your procedural sedation experience. After discharge patients will be contacted by phone 24 to 48 hours later to review a final questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I and II patients between the ages of 16 to 50 years scheduled to have their third molars extracted under intravenous sedation.

Exclusion Criteria:

* history of psychiatric illness, chronic use of central nervous system depressants or antidepressants, or alcohol abuse, had an active infection with systemic symptoms, were morbidly obese, were pregnant, or had a positive history of anesthetic-related complications.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 169 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pre-Sedation Behavioral Sate | Pre-operative assessment by RN the day of surgery just prior to entering the operating room.
  Patient will complete Corah anxiety scale.
Efficacy of Sedation | Monitored using a post-operative questionnaire administered 30 minutes after arrival to the recovery room.
  The patient does not have unpleasant recall of the procedure.
Adverse outcome | Throughout the procedural sedation in a continuous fashion. The start time of the procedural sedation will be defined as the time of the first dose of propofol and the stop time will be the time that the patient is transferred to recovery.
  Patient will be monitored for: apnea, aspiration, vomiting, cardiovascular events, excitatory movements, paradoxical response
Adverse outcomes | The patient will be monitored the recovery room in a continuous fashion for 30 minutes.
  Unpleasant recovery reactions, permanent complications.
Patient Satisfaction | This will be measured 30 minutes after arrival to the recovery room and then once again via phone questionnaire between 24 to 48 hours after discharge.
  A questionnaire will be given to the patient to complete just prior to discharge. The patient will be contacted 24 to 48 hours after discharge to complete a second questionnaire.
Level of sedation | This will be measured every 5 minutes throughout the duration of the procedural sedation.
  The Ramsay sedation scale will be used to grade the depth of sedation during the procedure.
Surgeon satisfaction | Immediately after completing the surgical procedure.
  The surgeon will complete a 5 point likert scale to determine their level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Davis, DDS FRCD(C), Principal Investigator — Staff Surgeon at "Atlantic Centre for Oral and Maxillofacial Surgery"
Locations (1):
- Atlantic Centre for Oral and Maxillofacial Surgery 1278 Tower Rd., Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Zed PJ, Abu-Laban RB, Chan WW, Harrison DW. Efficacy, safety and patient satisfaction of propofol for procedural sedation and analgesia in the emergency department: a prospective study. CJEM. 2007 Nov;9(6):421-7. doi: 10.1017/s148180350001544x. PMID 18072987
- [Result] Miner JR, Gray RO, Stephens D, Biros MH. Randomized clinical trial of propofol with and without alfentanil for deep procedural sedation in the emergency department. Acad Emerg Med. 2009 Sep;16(9):825-34. doi: 10.1111/j.1553-2712.2009.00487.x. PMID 19845550